CLINICAL TRIAL: NCT05113381
Title: A Prospective, Multicenter Study to Evaluate the Performance and Safety of the CerebroFlo™ EVD Catheter
Brief Title: The Purpose of This Study is to Determine Whether CerebroFlo™ EVD Catheter is Effective During the Treatment of Intraventricular Hemorrhage (IVH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-CERFLO-001
Record Dates: First submitted 2021-07-27; First posted 2021-11-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Intraventricular Hemorrhage; Subarachnoid Hemorrhage
Keywords: interventricular hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intraventricular Hemorrhage Subjects (Experimental): Intervention: Cerebrospinal Fluid (CSF) reduction Extra Ventricular Drainage (EVD) catheters will be used for cerebrospinal fluid drainage
  Interventions: Device: CerebroFlo™ EVD Catheter

INTERVENTIONS:
Device: CerebroFlo™ EVD Catheter — The CerebroFlo™ EVD Catheter is indicated for temporary insertion into a ventricular cavity of the brain for external drainage of cerebrospinal fluid (CSF) in those patients with elevated intracranial pressure (ICP), intraventricular hemorrhage, or hydrocephalic shunt infections.

SUMMARY:
The primary goal of this study is to assess the occurrence of flushing interventions to address occlusions during the treatment of interventricular hemorrhage (spontaneous primary IVH or secondary IVH due to ruptured aneurysm).

DETAILED DESCRIPTION:
Potential study candidates will be screened for inclusion and exclusion criteria after informed consent has been provided by the Legally Acceptable Representative and/or the study candidate.

Once enrolled in the study, data will be collected from those subjects with elevated intracranial pressure (ICP), interventricular hemorrhage, or hydrocephalic shunt infections as a result of the use of the EVD catheter.

Pre-insertion and peri-removal CT scans and neurological assessment data will also be collected.

Data will be collected for subjects beginning from the time of hospital admission through discharge and followed by the 30 Day and 90 Day Follow up Visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and/or legally authorized representative has reviewed the Institutional Review Board (IRB)-approved consent form, has been properly consented per the protocol and has documented their consent to participate in the study by signing the IRB-approved consent form.
2. Subject is ≥ 18 years of age at the time of consent.
3. Subjects with intraventricular hemorrhage (spontaneous primary IVH or secondary IVH due to ruptured aneurysm) who have had CerebroFlo™ EVD Catheter(s) placed without complication.
4. Subjects who require only one EVD Catheter at initial admission

Exclusion Criteria:

1. Subjects with a scalp infection present.
2. Subjects with uncorrectable coagulopathy due to prior administration of anticoagulants at the time the CerebroFlo™ EVD Catheter(s) is placed.
3. Subjects known to have a bleeding diathesis.
4. Subjects in which the CerebroFlo™ EVD Catheter(s) is placed directly into a hematoma
5. Evidence of catheter-associated hemorrhage from insertion of the CerebroFlo EVD Catheter(s) on post-placement CT scan.
6. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of flushing interventions to address occlusions | study device implantation through study device removal
  The number of flushing interventions from initial catheter placement through catheter removal, an average of 10 days, to address occlusions.

SECONDARY OUTCOMES:
Change of hemorrhage volume | Device implantation through to 90-Day follow-up
  Change of hemorrhage volume as assessed on pre- and post-insertion of the CerebroFlo device as assessed on CT scan
Assessment of Glasgow Coma Score (GCS) | Device implantation through to 90-Day follow-up
  Assessment of Glasgow Coma Score (GCS) at Admission, Discharge, 30-Day and/or 90-Day timepoints
  The Glasgow Coma Scale is divided into three components which are scored separately: ocular response (assessment 1-4 points), motor response (assessment 1-6 points) verbal response (evaluation of 1-5 points).
  Scores for each component are added together to get the total that will range between a minimum of 3 points (which corresponds to a patient who does not open his eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a patient with open eyes, obeying orders and maintaining a consistent language).
  It has been considered that the GCS score between 15 and 13 points corresponds to a slight alteration of consciousness, a score of 12-9 points with moderate impairment and 8 points or less with a serious deterioration in level of consciousness.
Assessment of Modified Rankin Score (mRS) | Device implantation through to 90-Day follow-up
  Assessment of Modified Rankin Score (mRS) at Admission, Discharge, 30-Day and/or 90-Day timepoints
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. Lower scores correlate with less disability/dependence
Assessment of National Institute of Health Stroke Scale (NIHSS) | Device implantation through to 90-Day follow-up
  Assessment of National Institute of Health Stroke Scale (NIHSS) at Admission, Discharge, 30-Day and/or 90-Day timepoints
  NIH Stroke Scale/Score (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Grandhi, MD, Principal Investigator — University of Utah Health; Jason Marzuola, MSN, Study Director — Integra Life Sciences
Locations (10):
- United States (10):
  - Loma Linda University Health, Loma Linda, California
  - Stanford University, Palo Alto, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Wright State University/Premier Health, Dayton, Ohio
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Virginia Commonwealth University Department of Neurosurgery, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aten Q, Killeffer J, Seaver C, Reier L. Causes, Complications, and Costs Associated with External Ventricular Drainage Catheter Obstruction. World Neurosurg. 2020 Feb;134:501-506. doi: 10.1016/j.wneu.2019.10.105. Epub 2019 Oct 25. PMID 31669535
- [Background] Fargen KM, Hoh BL, Neal D, O'connor T, Rivera-Zengotita M, Murad GJ. The burden and risk factors of ventriculostomy occlusion in a high-volume cerebrovascular practice: results of an ongoing prospective database. J Neurosurg. 2016 Jun;124(6):1805-12. doi: 10.3171/2015.5.JNS15299. Epub 2015 Oct 30. PMID 26517777
- [Background] Crites L. Reducing Catheter-Related Complications with New Anti-thrombiogenic PICC. JAVA. 2015:20(4):256.